CLINICAL TRIAL: NCT06991114
Title: An Open-label Phase 2a Study to Evaluate the Safety and Efficacy of AlloNK®, an Allogeneic Cord Blood-derived NK Cell Therapy, in Combination With Rituximab in Relapsing Forms of B-cell Dependent Rheumatologic Diseases
Brief Title: AlloNK®, an Allogeneic Non-genetically Modified, Cord Blood-derived NK Cell Therapy, in Combination With Rituximab, Studied in Relapsing Forms of B-cell Dependent Rheumatologic Diseases.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-101-05
Record Dates: First submitted 2025-05-19; First posted 2025-05-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Refractory Rheumatoid Arthritis (RA); Idiopathic Inflammatory Myopathies (IIMs); Systemic Sclerosis (SSc); Rheumatoid Arthritis (RA; IIM; Myositis; Scleroderma; Sjogren Syndrome; Sjogrens Disease
Keywords: Refractory Rheumatoid Arthritis; AlloNK; Idiopathic Inflammatory Myopathies; Systemic Sclerosis; Sjögren's Disease; Refractory RA; Cell Therapy; Allogeneic NK Cells; Allogeneic Cell Therapy; non-genetically modified; rituximab; cord blood cells; ADCC enhancement; outpatient; community
MeSH Terms: conditions — Arthritis, Rheumatoid; Myositis; Scleroderma, Systemic; Scleroderma, Diffuse; Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Open label, single group design to establish safety and efficacy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AlloNK (Experimental): AlloNK, dosed after a conditioning regimen, combined with Rituximab.
  Interventions: Drug: Allogeneic NK Cells

INTERVENTIONS:
Drug: Allogeneic NK Cells — AlloNK, dosed after a conditioning regimen, combined with Rituximab.

SUMMARY:
A Basket Trial of Refractory Rheumatoid Arthritis (RA), Sjögren's Disease (SjD), Idiopathic Inflammatory Myopathies (IIMs) and Systemic Sclerosis (SSc) subjects to evaluate the safety and efficacy of AlloNK, a non-genetically modified allogeneic NK cell, in combination with rituximab.

DETAILED DESCRIPTION:
An open-label Phase 2a study to evaluate the safety and efficacy of AlloNK®, an allogeneic cord blood-derived NK cell therapy, in combination with rituximab in relapsing forms of B-cell dependent rheumatologic diseases.

AlloNK® (also known as AB-101) is a non-genetically modified, allogeneic, off-the-shelf, cryopreserved cord blood-derived NK cell therapy.

ELIGIBILITY:
For Subjects with Refractory Rheumatoid Arthritis (RA):

* Documented diagnosis of RA, meeting the 2010 ACR/EULAR classification criteria.
* Rheumatoid Factor (RF) or Anti Citrullinated Protein Antibody (ACPA) positive.
* High-sensitivity C-reactive protein (hs-CRP) > 3 mg/L or Erythrocyte Sedimentation Rate (ESR) > 28 mm/hr.
* Have had prior treatment for a period of at least 12 weeks with a biologic disease modifying anti-rheumatic drug and were deemed refractory by the treating physician.
* Minimum of six swollen joint counts (SJC) and six tender joint counts (TJC) according to joint assessment.

For subjects with Sjögren's Disease (SjD)

* Prior diagnosis of Primary SjD as per 2016 ACR/EULAR criteria with confirmatory diagnosis in the 24 weeks preceding screening.
* Total Clinical European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (clinESSDAI) > 6.
* Salivary Flow Rate > 0.1 mL/min on stimulation.

For subjects with Idiopathic Inflammatory Myopathies (IIMs)

* Presence of a positive autoantibody (ANA >1:80 or RNP or SSA/SSB or other myositis specific autoantibodies.
* Refractory IIM as defined by inadequate response/intolerance to at least 3 months of glucocorticoids and/or at least one other immunosuppressive.
* Muscle biopsy or muscle MRI to confirm IIM diagnosis, where applicable, within 12 months prior to enrollment.

For Subjects with Systemic Sclerosis (SSc)

* Diagnosis of SSc in accordance with the ACR/EULAR 2013 classification.
* Modified Rodnan skin score (mRSS) > 10.
* Initial confirmatory diagnosis within 8 years of screening.
* Refractory SSc as defined by inadequate response/intolerance to at least 3 months of glucocorticoids and/or at least one other immunosuppressive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Safety | From enrollment until the end of treatment at Week 104.
  Dose Limiting toxicities assessed in a incrementing dose design.

SECONDARY OUTCOMES:
Rheumatoid Arthritis: Disease Activity Score 28 (DAS28 - ESR) | Week 52
  Efficacy
Sjögren's Disease: Improvement in Clinical EULAR Sjögren's Syndrome Disease Activity Index (ClinESSDAI) | Week 52
  Efficacy
Idiopathic Inflammatory Myopathies: Total Improvement Score (TIS) | Week 52
  Efficacy
Systemic Sclerosis: Revised Composite Response Index in Systemic Sclerosis (rCRISS) | Week 52
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saddekni, M.D., PgDip, BCMAS, Study Director — Artiva Therapeutics
Locations (25):
- United States (15):
  - Artiva Investigational Site Tuscaloosa, Tuscaloosa, Alabama
  - Artiva Investigational Site Phoenix, Phoenix, Arizona
  - Artiva Investigational Site Covina, Covina, California
  - Artiva Investigational Site Los Alamitos, Los Alamitos, California
  - Artiva Investigational Site Aventura, Aventura, Florida
  - Artiva Investigational Site Jupiter, Jupiter, Florida
  - Artiva Investigational Site Plantation, Plantation, Florida
  - Artiva Investigational Site Willowbrook, Willowbrook, Illinois
  - Artiva Investigational Site Iowa, Iowa City, Iowa
  - Artiva Investigational Site Charlotte, Charlotte, North Carolina
  - Artiva Investigational Site Hixson, Hixson, Tennessee
  - Artiva Investigational Site Arlington, Arlington, Texas
  - Artiva Investigational Site Katy, Katy, Texas
  - Artiva Investigational Site Mesquite, Mesquite, Texas
  - Artiva Investigational Site Woodland, Woodland, Texas
- Artiva Investigational Site Sofia, Sofia, Bulgaria
- France (3):
  - Artiva Investigational Site Marseille, Marseille
  - Artiva Investigational Site Montpellier, Montpellier
  - Artiva Investigational Site Toulouse, Toulouse
- Artiva Investigational Site Munchen, München, Germany
- Artiva Investigational Site Brescia, Brescia, Italy
- Artiva Investigational Site Vila Nova De Gaia, Vila Nova de Gaia, Portugal
- Romania (2):
  - Artiva Investigational Site Bucuresti, Bucharest
  - Artiva Investigational Site Bucharest, Bucharest
- Artiva Investigational Site Sevila, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided
AlloNK is early in clinical development, next steps will be based on the progress of our data.

REFERENCES:
- See also: Artiva AlloNK Basket Trial site. — https://allonk.patientwing.com/trials